CLINICAL TRIAL: NCT05036616
Title: Separation Versus Integrated Approach in Combining ECMO With CRRT, a Randomized Controlled Trial
Brief Title: Separation Versus Integrated Approach in Combining ECMO With CRRT
Acronym: E-CRRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Nattachai Srisawat ,M.D., Faculty of Medicine, Chulalongkorn University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB.151/64
Record Dates: First submitted 2021-08-26; First posted 2021-09-05 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: AKI
Keywords: CRRT; ECMO; integration; circuit; combination
MeSH Terms: interventions — Continuous Renal Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Separation technique (Experimental)
  Interventions: Device: Combination of extracorporeal membrane oxygenation and continuous renal replacement therapy
- Integration technique (Experimental)
  Interventions: Device: Combination of extracorporeal membrane oxygenation and continuous renal replacement therapy

INTERVENTIONS:
Device: Combination of extracorporeal membrane oxygenation and continuous renal replacement therapy — Combination of extracorporeal membrane oxygenation and continuous renal replacement therapy

SUMMARY:
This study aimed to compare circuit lifespan of CRRT between Integration and Separation techniques during ECMO support.

ELIGIBILITY:
ECMO patients >18 years old who met the KDIGO criteria for acute kidney injury and required continuous renal replacement therapy (CRRT). Inclusion criteria were as follows:

1. Refractory acidosis, defined as pH < 7.2 or serum bicarbonate (HCO₃-) < 15 mmol/L
2. Refractory volume overload
3. Refractory hyperkalemia, defined as serum potassium (K⁺) > 6.2 mEq/L or presence of electrocardiographic changes
4. Anuria or oliguria, defined as urine output < 0.5 mL/kg/hr for 6-12 hours
5. Elevated BUN >100 mg/dL or presence of uremic symptoms Increased intracranial pressure

Exclusion Criteria:

1. Pregnancy
2. Heparin contraindication
3. Chronic kidney disease with CRRT
4. AKI with Glomerulonephritis, Interstitial nephritis, Vassculitis or Urinary tract obstruction

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
CRRT Circuit lifespan | 72 hours, extended maximum to 120 hours
  The time until a CVVHDF malfunction was identified

SECONDARY OUTCOMES:
Serious Adverse Events | [Time Frame: 72 hours, extended maximum to 120 hours of filter lifespan]
  Bleeding at exit site, systemic bleeding, need for blood transfusion, air embolism, positive-blood culture infection, hemolysis
28-day mortality | 28-day after randomization
  28-day mortality, status yes or no
Pressure at various points of CRRT circuit | [Time Frame: 72 hours, extended maximum to 120 hours of filter lifespan]
  Pressure point at CRRT circuit; access pressure, return pressure, filter pressure, Pressure drop, and Transmembrane pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Sasipha tachaboon, Bangkok, Bangkok, Thailand

REFERENCES:
- [Background] Thy M, Augustin P, Tran-Dinh A, Montravers P, de Tymowski C. Renal Replacement Therapy for Patients Requiring Extracorporeal Membrane Oxygenation: A Multicenter International Survey. Blood Purif. 2022;51(11):899-906. doi: 10.1159/000522398. Epub 2022 Apr 7. PMID 35390796
- [Background] de Tymowski C, Desmard M, Lortat-Jacob B, Pellenc Q, Alkhoder S, Alouache A, Fritz B, Montravers P, Augustin P. Impact of connecting continuous renal replacement therapy to the extracorporeal membrane oxygenation circuit. Anaesth Crit Care Pain Med. 2018 Dec;37(6):557-564. doi: 10.1016/j.accpm.2018.02.024. Epub 2018 Mar 20. PMID 29572101
- [Derived] Tangjitaree P, Thanapongsatorn P, Sinjira T, Surinrat E, Suttiruk P, Srisawat N. The comparison of circuit lifespan between integration and separation approach in extracorporeal membrane oxygenation patients requiring continuous renal replacement therapy support: a randomized controlled trial (E-CRRT Trial). Intensive Care Med. 2026 Feb 5. doi: 10.1007/s00134-026-08302-y. Online ahead of print. PMID 41642325